CLINICAL TRIAL: NCT06560502
Title: A Multicenter, Prospective, Randomized Controlled Modified Multi-Platform (Matriarch) Trial Evaluating Several Cellular, Acellular, and Matrix-like Products (CAMPs) and Standard of Care Versus Standard of Care Alone in the Management of DFUs and VLUs.
Brief Title: Modified Multi-Platform Trial Assessing Multiple CAMPs and SOC vs SOC Alone in the Treatment of DFU and VLUs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stability Biologics (Industry)
Collaborators: SerenaGroup, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STABLECAMP
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Diabetic Foot Ulcer; Venous Leg Ulcer; Ulcer Foot; Leg Ulcer
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer; Foot Ulcer; Leg Ulcer

STUDY DESIGN:
Intervention Model Description: The study design is a prospective modified dual platform (matriarch) multicenter randomized controlled clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Standard of Care-DFU (Active Comparator): Debridement, reduction of bacterial burden, and proper moisture balance using dressings provided by SerenaGroup. Off-loading using the off-loading boot or total contact cast (TCC) provided by SerenaGroup.
  Interventions: Other: Standard of Care-DFU
- AmnioCore - DFU (Experimental): Dual layer, amniotic membrane allograft.
  Interventions: Other: AmnioCore - DFU
- Amnio Quad-Core - DFU (Experimental): Four layer, amniotic membrane allograft.
  Interventions: Other: Amnio Quad-Core - DFU
- Amniocore Pro + - DFU (Experimental): Dual layer, amnion/chorion membrane allograft.
  Interventions: Other: Amniocore Pro +
- Standard of Care-VLU (Active Comparator): Debridement, reduction of bacterial burden, and proper moisture balance using dressings provided by SerenaGroup. Compression using multilayer compression wraps provided by SerenaGroup.
  Interventions: Other: Standard of Care-VLU
- Amnio Tri-Core - VLU (Experimental): Three layer, amniotic membrane allograft.
  Interventions: Other: Amnio Tri-Core - VLU
- AmnioCore Pro - VLU (Experimental): Three layer, amnion/chorion/amnion membrane allograft.
  Interventions: Other: AmnioCore Pro

INTERVENTIONS:
Other: Standard of Care-DFU — Beginning at the screening visit, participants will receive weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and offloading) until ulcer closure, or a maximum of 13 weeks, whichever occurs first.
  Arms: Standard of Care-DFU
Other: AmnioCore - DFU — Participants will receive weekly applications of AmnioCore and Standard of Care until ulcer closure, or a maximum of 13 weeks, whichever occurs first.
  Arms: AmnioCore - DFU
Other: Amnio Quad-Core - DFU — Participants will receive weekly applications of Amnio Quad-Core and Standard of Care until ulcer closure, or a maximum of 13 weeks, whichever occurs first.
  Arms: Amnio Quad-Core - DFU
Other: Standard of Care-VLU — Beginning at the screening visit, participants will receive weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and compression) until ulcer closure, or a maximum of 13 weeks, whichever occurs first.
  Arms: Standard of Care-VLU
Other: Amnio Tri-Core - VLU — Participants will receive weekly applications of Amnio Tri-Core and Standard of Care until ulcer closure, or a maximum of 13 weeks, whichever occurs first.
  Arms: Amnio Tri-Core - VLU
Other: AmnioCore Pro — Participants will receive weekly applications of AmnioCore Pro and Standard of Care until ulcer closure, or a maximum of 13 weeks, whichever occurs first.
  Arms: AmnioCore Pro - VLU
Other: Amniocore Pro + — Participants will receive weekly applications of Amniocore Pro + and Standard of Care until ulcer closure, or a maximum of 13 weeks, whichever occurs first.
  Arms: Amniocore Pro + - DFU

SUMMARY:
This is a multicenter, prospective, randomized controlled modified multi-platform (matriarch) trial evaluating several cellular, acellular, and matrix-like products (CAMPs) and standard of care versus standard of care alone in the management of nonhealing diabetic foot and venous leg ulcers.

DETAILED DESCRIPTION:
The purpose of this study is to determine the between-arm difference in the proportion of subjects achieving complete closure of nonhealing diabetic foot ulcers and venous leg ulcers with multiple CAMPs plus SOC versus SOC alone over 12 weeks using a modified dual platform (Matriarch) trial design.

*The initial plan is to evaluate five CAMPs per wound type; however, the modified platform design permits the inclusion of additional CAMPs.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects must be at least 21 years of age or older. 2. Subjects must have a diagnosis of type 1 or 2 Diabetes mellitus. 3. At randomization subjects must have a target ulcer with a minimum surface area of 1.0 cm2 and a maximum surface area of 5.0 cm2 measured post debridement .

  4. The target ulcer must have been present for a minimum of 4 weeks and a maximum of 52 weeks of standard of care, prior to the initial screening visit.

  5. The target ulcer must be located on the foot with at least 50% of the ulcer below the malleolus.

  6. The target ulcer must be Wagner 1 or 2 grade, extending at least through the dermis or subcutaneous tissue and may involve the muscle provided it is below the medial aspect of the malleolus.

  7. The affected limb must have adequate perfusion confirmed by vascular assessment. Any of the following methods performed within 3 months of the first screening visit are acceptable:

  a. ABI between 0.7 and ≤ 1.3; b. TBI ≥ 0.6; c. TCOM ≥ 40 mmHg; d. PVR: biphasic. 8. If the potential subject has two or more ulcers, they must be separated by at least 2 cm post-debridement. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer.

  9. Target ulcers located on the plantar aspect of the foot must be offloaded for at least 14 days prior to enrollment.

  10. The potential subject must consent to using the prescribed offloading method for the duration of the study.

  11. The potential subject must agree to attend the weekly study visits required by the protocol.

  12. The potential subject must be willing and able to participate in the informed consent process.

Exclusion Criteria:

1. The potential subject is known to have a life expectancy of < 6 months.
2. The potential subject's target ulcer is not secondary to diabetes.
3. The target ulcer is infected, requires systemic antibiotic therapy, or there is cellulitis in the surrounding skin.
4. The target ulcer exposes tendon or bone.
5. There is evidence of osteomyelitis complicating the target ulcer.
6. The potential subject is receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of prednisone per day or equivalent) or cytotoxic chemotherapy or is taking medications that the PI believes will interfere with wound healing (e.g., biologics).
7. The potential subject is taking hydroxyurea .
8. The potential subject has applied topical steroids to the ulcer surface within one month of initial screening.
9. The potential subject with a previous partial amputation on the affected foot that results in a deformity that impedes proper offloading of the target ulcer.
10. The potential subject has glycated hemoglobin (HbA1c) greater than or equal to 12% within 3 months of the initial screening visit.
11. The surface area of the target ulcer has reduced in size by more than 20% in the 2 weeks prior to the initial screening visit ("historical" run-in period). MolecuLight Imaging Device is not required for measurements taken during the historical run-in period (e.g., calculating surface area using length X width is acceptable).
12. The surface area measurement of the Target ulcer decreases by 20% or more during the active 2-week screening phase: the 2 weeks from the initial screening visit (SV-1) to the TV-1 visit during which time the potential subject received SOC.
13. The potential subject has an acute Charcot foot, or an inactive Charcot foot, which impedes proper offloading of the target ulcer.
14. Women who are pregnant or considering becoming pregnant within the next 6 months.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Determine the between-arm difference | 1-12 Weeks
  To determine the between-arm difference in the proportion of subjects achieving complete closure of nonhealing diabetic foot ulcers and venous leg ulcers with multiple CAMPs plus SOC versus SOC alone over 12 weeks using a modified dual platform (Matriarch) trial design.

SECONDARY OUTCOMES:
Time to closure | 1-12 Weeks
  To determine the between-arm difference in the time to closure over 12 weeks for CAMP plus SOC versus SOC alone.
Percent Area Reduction | 1-12 weeks
  To determine the between-arm difference in the percent area reduction (PAR) at weekly intervals the CAMP plus SOC arms versus SOC alone.
Change in pain in target ulcer | 1-12 Weeks
  To determine the between-arm difference in pain for patients that present with a VAS score of greater than 4.
Adverse Events | 1-14 weeks
  To evaluate the between-arm difference in the frequency and nature of adverse events in subjects receiving CAMP plus SOC versus SOC alone.
Determine improvement in Quality of Life - FWS and determine improvement in Quality of Life - wQOL | 1-12 weeks
  To evaluate the between-arm difference in the quality of life for subjects receiving CAMP plus SOC compared to SOC alone using the Forgotten Wound Score (FWS) and standard Wound Quality of Life (wQOL) questionnaires at treatment visits 1, 4, 8, and 12.

CONTACTS AND LOCATIONS:
Locations (1):
- Cutting Edge Research, Circleville, Ohio, United States

IPD SHARING:
Plan to Share IPD: No